CLINICAL TRIAL: NCT02659592
Title: Transplantation of Frozen Thawed Ovarian Tissue Demonstrates High Reproductive Performance and the Need to Revise Restrictive Criteria
Brief Title: Transplantation of Frozen Thawed Ovarian Tissue High Reproductive Performance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Dror Meirow, professor, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-03-3026-DM-CTIL
Record Dates: First submitted 2016-01-07; First posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Reproductive Performance Following Ovarian Transplantation
Keywords: fertility preservation; ovarian tissue transplantation; ovarian endocrine function; assisted reproductive technology; pregnancy and live birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- infertile cancer survivors (Experimental): infertile cancer survivors who seek to conceive and had frozen ovarian tissue when diagnosed years before
  Interventions: Procedure: transplantation of ovarian tissue

INTERVENTIONS:
Procedure: transplantation of ovarian tissue — operation(mini laparotomy) for transplantation of frozen- thawed ovarian tissue

SUMMARY:
Design: prospective cohort study. Setting: Tertiary university-affiliated ART and oncology centers. Patients: 20 cancer survivors who underwent ovarian transplantation of frozen-thawed ovarian tissue, with the aim to conceive.

Interventions: Ovarian tissue cryopreservation (OTCP) and transplantation, endocrine monitoring, IVF.

DETAILED DESCRIPTION:
Main Outcomes expected:

Endocrine profile IVF results, pregnancy rates following transplantation of ovarian tissue live-births rates following transplantation of ovarian tissue cancer disease recurrence

ELIGIBILITY:
Inclusion Criteria: infertile patients who stored ovarian tissue to preserve fertility prior to potentially sterilizing cancer treatments

-

Exclusion Criteria:

* active disease, fertile patients post cancer treatment

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-01; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
menstrual bleeding (yes/no) | up to one year
  recurrence of menstrual bleeding- yes or no
number of oocytes per IVF cycle | through study completion (up to 11 years following transplantation)
  number of aspirated oovytes per one IVF cycle performed
pregnancies | through study completion (up to 11 years following transplantation)
  spontaneous or post IVF pregnancy rates (%)
live births | through study completion (up to 11 years following transplantation)
  live birth rates (%)

SECONDARY OUTCOMES:
disease reccurence | through study completion (7 months to 141 months following transplantation)
  incidence of cancer disease recurrence

OTHER OUTCOMES:
FSH levels (miU/ml) | up to one year
  as part of the endocrine profile
E2 (pmol/ml), | up to one year
  as part of the endocrine profile
number of embryos per IVF cycle | through study completion (up to 11 years following transplantation)
IVF cycles pregnancy rates (%) | through study completion (up to 11 years following transplantation)
  number of pregnancies obtained via IVF devided by number of IVF cycles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meirow D, Ra'anani H, Shapira M, Brenghausen M, Derech Chaim S, Aviel-Ronen S, Amariglio N, Schiff E, Orvieto R, Dor J. Transplantations of frozen-thawed ovarian tissue demonstrate high reproductive performance and the need to revise restrictive criteria. Fertil Steril. 2016 Aug;106(2):467-74. doi: 10.1016/j.fertnstert.2016.04.031. Epub 2016 May 12. PMID 27181924